CLINICAL TRIAL: NCT02051816
Title: Facilitating EndotracheaL Intubation by Laryngoscopy Technique and Apneic Oxygenation Within the Intensive Care Unit
Brief Title: Facilitating EndotracheaL Intubation by Laryngoscopy Technique and Apneic Oxygenation Within the Intensive Care Unit: The FELLOW Study
Acronym: FELLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, David Janz, Clinical Fellow, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 131966
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Respiratory Failure
Keywords: Endotracheal Intubation; Apneic Oxygenation; Respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- VL and AO (Active Comparator): Video laryngoscopy and apneic oxygenation
  Interventions: Device: Apneic Oxygenation; Device: No Apneic Oxygenation
- DL and AO (Active Comparator): Direct Laryngoscopy and apneic oxygenation
  Interventions: Device: Apneic Oxygenation; Device: No Apneic Oxygenation
- VL and no AO (Active Comparator): Video Laryngoscopy and no apneic oxygenation
  Interventions: Device: Video Laryngoscopy; Device: Direct Laryngoscopy
- DL and no AO (Active Comparator): Direct Laryngoscopy and no apneic oxygenation
  Interventions: Device: Video Laryngoscopy; Device: Direct Laryngoscopy

INTERVENTIONS:
Device: Video Laryngoscopy
  Arms: DL and no AO; VL and no AO
Device: Apneic Oxygenation
  Arms: DL and AO; VL and AO
Device: Direct Laryngoscopy
  Arms: DL and no AO; VL and no AO
Device: No Apneic Oxygenation
  Arms: DL and AO; VL and AO

SUMMARY:
Respiratory failure requiring endotracheal intubation occurs in as many as 40% of critically ill patients. Procedural complications including failed attempts at intubation, esophageal intubation, arterial oxygen desaturation, aspiration, hypotension, cardiac arrest, and death are common in this setting. While there are many important components of successful airway management in critical illness, the maintenance of adequate arterial hemoglobin saturation from procedure initiation until endotracheal tube placement is paramount as desaturation is the most common factor associated with peri-intubation cardiac arrest and death. Interventions that either shorten the duration of time required for tube placement or prolong the period before desaturation may be effective in improving outcome. The high rate of complications and the lack of existing evidence regarding the efficacy of current airway management techniques in shortening the time to airway establishment or prolonging the time to desaturation mandates further investigation. The primary hypothesis is that video laryngoscopy will be superior to direct laryngoscopy in successful first attempt at endotracheal intubation (defined by confirmed placement of an endotracheal tube in the trachea during first laryngoscopy attempt) of medical ICU patients by Pulmonary/Critical Care Medicine fellows after controlling for the operator's past number of procedures with the equipment used. Also, the investigators hypothesize that the provision of apneic oxygenation during the endotracheal intubation procedure (defined as a nasal cannula with 15 liters per minute of oxygen flow placed prior to sedation or neuromuscular blockade and maintained until after completion of the procedure) will result in a higher arterial oxygen saturation nadir (defined as lowest noninvasive oxygenation saturation value observed between the administration of sedation and/or neuromuscular blockade and 2 minutes after successfully secured airway or death) compared to no apneic oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Medical ICU Patients
* Require endotracheal intubation
* Endotracheal intubation to be performed by Pulmonary/Critical Care Medicine Fellow
* Sedation and/or neuromuscular blockade is planned for the procedure

Exclusion Criteria:

* Operators other than Pulmonary/Critical Care Medicine Fellows
* The operator predetermines that the patient requires specific intubating equipment or oxygenation technique will be required for the safe performance of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Semler, MD, Principal Investigator — Vanderbilt University; Todd W Rice, MD, MSc, Study Chair — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Semler MW, Janz DR, Lentz RJ, Matthews DT, Norman BC, Assad TR, Keriwala RD, Ferrell BA, Noto MJ, McKown AC, Kocurek EG, Warren MA, Huerta LE, Rice TW; FELLOW Investigators; Pragmatic Critical Care Research Group. Randomized Trial of Apneic Oxygenation during Endotracheal Intubation of the Critically Ill. Am J Respir Crit Care Med. 2016 Feb 1;193(3):273-80. doi: 10.1164/rccm.201507-1294OC. PMID 26426458

RESULTS

PARTICIPANT FLOW:
Groups:
- Video Laryngoscopy and No Apneic Oxygenation: Patients randomized to undergo endotracheal intubation using the operator's choice of McGrath® video laryngoscope, GlideScope® video laryngoscope, or bronchoscope.
  No Apneic Oxygenation
- Direct Laryngoscopy and Apneic Oxygenation: Patients randomized to undergo endotracheal intubation using the operator's choice of a MacIntosh or Miller blade direct laryngoscope.
  Apneic Oxygenation
- Video Laryngoscopy and Apneic Oxygenation: A nasal cannula with 15 liters per minute of oxygen flow placed prior to sedation or neuromuscular blockade and maintained until after completion of the procedure
  Video Laryngoscopy
- Direct Laryngoscopy and No Apneic Oxygenation: No nasal cannula, supplemental oxygen given after sedation or neuromuscular blockade until completion of the procedure.
  Direct Laryngoscopy
Period: Overall Study
Arm/Group | Video Laryngoscopy and No Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation
Started | 37 | 40 | 37 | 36
Completed | 37 | 40 | 37 | 36
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Video Laryngoscopy and Apneic Oxygenation: Patients randomized to undergo endotracheal intubation using the operator's choice of McGrath® video laryngoscope, GlideScope® video laryngoscope, or bronchoscope.
  and
  A nasal cannula with 15 liters per minute of oxygen flow placed prior to sedation or neuromuscular blockade and maintained until after completion of the procedure
- Direct Laryngoscopy and Apneic Oxygenation: Patients randomized to undergo endotracheal intubation using the operator's choice of a MacIntosh or Miller blade direct laryngoscope.
  and
  A nasal cannula with 15 liters per minute of oxygen flow placed prior to sedation or neuromuscular blockade and maintained until after completion of the procedure
- Video Laryngoscopy and no Apneic Oxygenation: Patients randomized to undergo endotracheal intubation using the operator's choice of McGrath® video laryngoscope, GlideScope® video laryngoscope, or bronchoscope.
  and
  No apneic oxygenation
- Direct Laryngoscopy and No Apneic Oxygenation: Patients randomized to undergo endotracheal intubation using the operator's choice of a MacIntosh or Miller blade direct laryngoscope.
  and
  No apneic oxygenation
- Total: Total of all reporting groups
Arm/Group | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and no Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation | Total
Number analyzed (Participants) | 37 | 40 | 37 | 36 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (15) | 58 (14) | 56 (15) | 58 (12) | 58 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 12 | 15 | 59
  Male | 22 | 23 | 25 | 21 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 6 | 3 | 19
  White | 33 | 30 | 30 | 32 | 125
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 1 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 37 | 40 | 37 | 36 | 150
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29 (8) | 29 (9) | 28 (5) | 29 (8) | 29 (8)
Acute Physiology and Chronic Health Evaluation II Score [Mean (Standard Deviation); unit: units on a scale] — range of scale is minimum 0 - maximum 100 lower values describe less acute/chronic illness and more likely to survive higher values describe more acute/chronic illness and less likely to survive
  units on a scale | 21 (9) | 21 (6) | 23 (6) | 21 (6) | 21 (7)

OUTCOME MEASURES:

1. Primary Outcome: Successful First Attempt at Endotracheal Intubation (Defined by Confirmed Placement of an Endotracheal Tube in the Trachea During First Laryngoscopy Attempt) After Controlling for the Operator's Past Number of Procedures With the Equipment Used.
Description: The primary outcome for the video laryngoscopy compared with direct laryngoscopy arm of the study will be the successful first attempt at endotracheal intubation (defined by confirmed placement of an endotracheal tube in the trachea during first laryngoscopy attempt) after controlling for the operator's past number of procedures with the equipment used.
Time Frame: 1 hour
Measure: Number; unit: participants
Groups:
- Video Laryngoscopy: Patients randomized to undergo endotracheal intubation using the operator's choice of McGrath® video laryngoscope, GlideScope® video laryngoscope, or bronchoscope.
  Apneic Oxygenation
  No Apneic Oxygenation
- Direct Laryngoscopy: Patients randomized to undergo endotracheal intubation using the operator's choice of a MacIntosh or Miller blade direct laryngoscope.
  Apneic Oxygenation
  No Apneic Oxygenation
- Apneic Oxygenation: A nasal cannula with 15 liters per minute of oxygen flow placed prior to sedation or neuromuscular blockade and maintained until after completion of the procedure
  Video Laryngoscopy
  Direct Laryngoscopy
- No Apneic Oxygenation: No nasal cannula, supplemental oxygen given after sedation or neuromuscular blockade until completion of the procedure.
  Video Laryngoscopy
  Direct Laryngoscopy
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy | Apneic Oxygenation | No Apneic Oxygenation
Number analyzed (Participants) | 74 | 76 | 77 | 73
participants | 51 | 50 | NA — See apneic oxygenation separate outcomes | NA — See apneic oxygenation separate outcomes

2. Primary Outcome: Arterial Oxygen Saturation Nadir (Defined as Lowest Noninvasive Oxygenation Saturation Value Observed Between the Administration of Sedation and/or Neuromuscular Blockade and 2 Minutes After Successfully Secured Airway or Death).
Description: The primary outcome for the apneic oxygenation arm of the study is arterial oxygen saturation nadir (defined as lowest noninvasive oxygenation saturation value observed between the administration of sedation and/or neuromuscular blockade and 2 minutes after successfully secured airway or death).
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: percent arterial oxygen saturation
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy | Apneic Oxygenation | No Apneic Oxygenation
Number analyzed (Participants) | 74 | 76 | 77 | 73
percent arterial oxygen saturation | NA [NA to NA] — See video laryngoscopy outcomes separately | NA [NA to NA] — See video laryngoscopy outcomes separately | 92 [84 to 99] | 90 [80 to 96]

3. Secondary Outcome: Procedure-related Mortality
Description: Death within 1 hour of beginning the procedure
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscopy and No Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation
Number analyzed (Participants) | 37 | 40 | 37 | 36
Participants | 0 | 0 | 0 | 1

4. Secondary Outcome: ICU-mortality
Description: Death from any cause in the ICU and at anytime after the procedure
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscopy and No Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation
Number analyzed (Participants) | 37 | 40 | 37 | 36
Participants | 19 | 15 | 12 | 17

5. Secondary Outcome: Adjusted Lowest Arterial Oxygen Saturation During Procedure
Description: Arterial oxygen saturation nadir (defined as lowest noninvasive oxygenation saturation value observed between the administration of sedation and/or neuromuscular blockade and 2 minutes after successfully secured airway or death) adjusted for arterial oxygen saturation at the time of administering intubation drugs.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: PERCENT SATURATION
Arm/Group | Video Laryngoscopy and No Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation
Number analyzed (Participants) | 37 | 40 | 37 | 36
PERCENT SATURATION | 88 (12) | 89 (12) | 87 (12) | 82 (16)

6. Secondary Outcome: Ventilator-free Days
Description: Number of days alive and free of mechanical ventilation after endotracheal intubation
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: DAYS
Arm/Group | Video Laryngoscopy and No Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation
Number analyzed (Participants) | 37 | 40 | 37 | 36
DAYS | 9 (12) | 12 (12) | 14 (12) | 11 (12)

7. Secondary Outcome: Number of Esophageal Intubations Per Group
Description: Number of esophageal intubations Per Study Group
Time Frame: 1 hour
Measure: Number; unit: number of esophageal intubations
Arm/Group | Video Laryngoscopy and No Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation
Number analyzed (Participants) | 37 | 40 | 37 | 36
number of esophageal intubations | 0 | 1 | 1 | 3

8. Secondary Outcome: Grade View of the Glottis
Description: Best Cormack-Lehane grade view of the glottis (grade 1-4) on first laryngoscopy attempt. Higher grades on the 1-4 scale indicate worse glottic views.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video Laryngoscopy and No Apneic Oxygenation | Direct Laryngoscopy and Apneic Oxygenation | Video Laryngoscopy and Apneic Oxygenation | Direct Laryngoscopy and No Apneic Oxygenation
Number analyzed (Participants) | 37 | 40 | 37 | 36
units on a scale | 1.24 (.43) | 1.8 (1.09) | 1.3 (.66) | 1.75 (.77)

ADVERSE EVENTS:
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy | Apneic Oxygenation | No Apneic Oxygenation
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76 | 0/77 | 0/73
Other Adverse Events (participants affected / at risk) | 0/74 | 0/76 | 0/77 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No